CLINICAL TRIAL: NCT04932837
Title: Determination of the Level of Immunity, Neutralization of the SARS-COV-2 Virus and Reinfections in Residents of 2 Migrant Workers' Residences 10 Months Apart
Brief Title: Level of Immunity, Neutralization of the COVID-19 Virus and Reinfections in Residents of 2 Migrant Workers' Residences
Status: Withdrawn | Type: Observational
Why Stopped: The vaccination campaign started before the approval of the ethics committee was obtained. The study is therefore no longer of interest to be carried out.
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); Institut Pasteur (Industry); Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 811562
Record Dates: First submitted 2021-06-01; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: SARS-COV-2
Keywords: COVID-19; migrant workers' residences; Immunity; protection
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- migrant worker residents: The target population will be the 124 residents in the 2 migrant worker residences who were included in the previous seroprevalence study and those who arrived at the 2 residences since September 1st, 2020
  Interventions: Biological: Blood and Saliva collection

INTERVENTIONS:
Biological: Blood and Saliva collection — Serological, viral RNA and antigenic test

SUMMARY:
A previous seroprevalence survey showed very high seroprevalence levels among residents of the two among the residents of the two migrant workers' hostels surveyed, indicating a high level of circulation of the virus SARS-COV-2 during the 1st wave of COVID-19. The constitution of a cohort after the event would be an opportunity to obtain opportunity to obtain answers to crucial questions: duration of immunity, potential reinfections potential reinfections, potential re-clustering. Going back to check the serological status seems feasible, especiallyespecially in the Foyers de Travailleurs Migrants (high probability of finding the participants).

There is an obvious scientific interest around the duration of immunity and reinfections in a population highly exposed during the first wave. Several articles document the decline of IgG antibodies in the months following an infection, but very few infection, but very few evaluate the protective character in the medium term (>=6 months), especially in asymptomatic individuals. We are also concerned about the circulation of We are also concerned about the circulation of new variants and the immunity acquired after infection in residents.

To date, no study on the duration of immunity has been conducted in migrant worker's residences.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who consented to participate in the 1st study and who consent to participate in this study
* All individuals 18 years of age or older not residing in the 2 MWRs in July 2020 and permanently living in the MWR since September 2020 who consent to participate in this study

Exclusion Criteria:

* Unwillingness to provide informed consent
* Unwillingness to provide blood
* Contraindication to venepuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of 2 Migrant Workers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-14 (Estimated); Primary Completion 2021-06-25 (Estimated); Study Completion 2021-07-02 (Estimated)

PRIMARY OUTCOMES:
Level and quality of current humoral immune protection in the residents of the two migrant workers' residences | 15 days
  To assess the level and quality of current humoral immune protection in the residents of the two migrant workers' residences in Villemomble and Montreuil who were included in the 1st seroprevalence study in July 2020, approximately 10 months later (May 2021)

SECONDARY OUTCOMES:
Immunity and protection | 15 days
  * Identify potential reinfections (reported symptoms confirmed by positive PCR tests) or resurgence of symptoms (long COVID) among residents who were seropositive in July 2020
  * Assess the evolution of antibodies (IgA, IgM, IgG) approximately 10 months after the first test in Sars-CoV-2 seropositive individuals in July
  * To evaluate the neutralizing and therefore protective activity of the re-measured antibodies, and their level of affinity maturation to SARS-COV-2 as well as their efficacy against the mainly circulating variants: B.1.1.7 (UK), B.1.351 (South Africa) and P.1 (Brazil)
New infections and screening | 15 days
  * Estimate the proportion of infections (reported symptoms and/or positive PCR tests)/exposure to the virus in people newly arrived since September 2020
  * In case of SARS-COV-2 RNA detection, characterize the virus subtype (genomic sequencing)
  * Document the turnover in MWR populations to guide MSF activities in the future
COVID Vaccination | 15 days
  * Assess the proportion of participants already vaccinated or interested in the future COVID vaccination campaign and document the reasons for those who express doubts or plan to refuse vaccination
  * To evaluate the performance of the LuLISA technique for the response to SARS-CoV-2 N and S proteins
  * To evaluate the performance of a rapid serological test on strip, LuLISA Stripe developed by the Institute Pasteur by comparison to the LuLISA technique
  * To evaluate the performance of a rapid N and S antigenic test on saliva, LuLISA Flash, developed by the Institut Pasteur, by comparing it to the RT-PCR method
  * To evaluate the performance of an alternative antigenic test on saliva with very high sensitivity, LuLISA Stick, developed by Institute Pasteur, by comparing it to the RT-PCR method
  * Evaluate the performance of a rapid molecular RT-LAMP test developed by Institute Pasteur (depending on availability) by comparing it to the RT-PCR method

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth POULET, MD, Principal Investigator — Epicentre
Locations (2):
- France (2):
  - Foyer de travailleurs migrants, Montreuil, Île-de-France Region
  - Foyer de travailleurs migrants, Villemomble, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The research team will develop a range of activities to disseminate the study findings. These dissemination activities will be coordinated by MSF and Epicentre. The results will be presented in an internal report and an external report for the Ministry of Health (MoH), the French National Public Health Agency and Institute Pasteur.
  An abstract of the findings will be submitted for presentation at a scientific conference, and at least one manuscript will be submitted for publication in a peer-reviewed scientific journal.
  The findings of the survey will also be used for advocacy purposes, in coordination with community leaders of participating communities.
  The results of the survey (lay version of the report), and their possible use for advocacy / communication, will be shared with the staff, resident representatives and residents of the MWRs, whether or not they actually participated in the study.
Supporting Information: CSR